CLINICAL TRIAL: NCT01582854
Title: A 12-month, International, Parallel Group, Randomised, Multi-centre, Double-blind, Placebo-controlled Trial to Examine the Effect of Actovegin® Treatment Given First Intravenously and Subsequently Orally Over 6 Months, in Subjects With Post-stroke Cognitive Impairment (PSCI).
Brief Title: Efficacy and Safety of Actovegin in Post-stroke Cognitive Impairment (PSCI)
Acronym: ARTEMIDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV-2500-301-RD; U1111-1132-3434 (Registry Identifier: WHO)
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Post-Stroke Cognitive Impairment (PSCI)
Keywords: Post-Stroke Cognitive Impairment (PSCI); Stroke; Actovegin; Cognition disorders
MeSH Terms: conditions — Stroke; Cognition Disorders | interventions — Actovegin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Actovegin (Active Comparator): Actovegin 2000 mg solution, intravenous (IV) infusion for up to 20 days followed by 2 actovegin 200 mg, tablets, orally, 3 times a day for up to 6 months.
  Interventions: Drug: Actovegin
- Placebo (Placebo Comparator): Actovegin placebo-matching solution, intravenous (IV) infusion for up to 20 days followed by 2 actovegin placebo-matching, tablets, orally, 3 times a day for up to 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Actovegin — Actovegin solution for infusion and Actovegin tablets
  Arms: Actovegin
Drug: Placebo — Actovegin placebo-matching solution for infusion and Actovegin placebo-matching tablets
  Arms: Placebo

SUMMARY:
The aim of this trial is to provide evidence that Actovegin has a symptomatic effect in subjects with post stroke cognitive impairment (PSCI) during a six month treatment period compared to subjects administered placebo. Subjects received IV infusions whilst in hospital, and tablets once discharged. Subjects were followed up for a further six months after their treatment had been stopped to explore if the cognitive symptoms of the subjects treated with Actovegin showed sustained improvement. The trial also explored the possible prevention of dementia with Actovegin in patients who had suffered a recent ischaemic stroke, as well as the effect of Actovegin on other stroke outcomes. Safety information on Actovegin was collected.

DETAILED DESCRIPTION:
The drug tested in this study is called actovegin. Actovegin was tested to treat people who have post stroke cognitive impairment. This study looked at the improvement of cognitive symptoms in people who take actovegin compared to placebo.

The study enrolled 503 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study:

* Actovegin-2000 mg intravenous solution; 2- 200 mg tablets 3 times a day
* Placebo intravenous solution; tablets (dummy inactive) - this is a solution or tablet that looks like the study drug but has no active ingredient

All participants received daily intravenous infusions in the hospital (up to a maximum of 20 infusions) followed by 2-200 mg tablets three times a day for the remainder of the 6-month treatment period.

This multi-centre trial was conducted in Belarus, Kazakhstan and Russia. The overall time to participate in this study was 12 months. Participants made multiple visits to the clinic plus a final visit after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant has suffered a recent supra-tentorial ischaemic stroke supported by computed tomography (CT) scan or magnetic resonance imaging (MRI) findings (in accordance with local practice).
* Participant is male or female, aged 60 years or above.
* Participant has a score on the National Institute of Health Stroke Scale (NIHSS) between 3 and 18 (inclusive).
* Participant is capable of completing the Montreal Cognitive Assessment (MoCA) and has a score of ≤ 25 points with adjustment for level of education (4-9 school years ≤ 23 points, 10-12 years ≤ 24 points, >12 years ≤ 25 points).

Main Exclusion Criteria:

* Participant has a medical history of dementia.
* Participant has a known medical history of major depression or psychotic disorder.
* Participant is indicated for treatment with thrombolytics or carotid surgery as the current standard of care.

Randomisation Criteria:

* Inclusion Criteria.
* Ability to perform Alzheimer's Disease Assessment Scale + Cognitive Subscale Extended Version (ADAS-cog+).
* Exclusion Criteria.
* Clinically there is suspicion of progressive stroke.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Belarus (3):
  - Nycomed Investigational Site, Grodno
  - Nycomed Investigational Site, Minsk
  - Nycomed Investigational Site, Vitebsk
- Nycomed Investigational Site, Almaty, Kazakhstan
- Russia (10):
  - Nycomed Investigational Site, Barnaul
  - Nycomed Investigational Site, Irkutsk
  - Nycomed Investigational Site, Kazan'
  - Nycomed Investigational Site, Krasnoyarsk
  - Nycomed Investigational Site, Moscow
  - Nycomed Investigational Site, Novosibirsk
  - Nycomed Investigational Site, Saint Petersburg
  - Nycomed Investigational Site, Samara
  - Nycomed Investigational Site, Tomsk
  - Nycomed Investigational Site, Yekaterinburg

REFERENCES:
- [Derived] Guekht A, Skoog I, Edmundson S, Zakharov V, Korczyn AD. ARTEMIDA Trial (A Randomized Trial of Efficacy, 12 Months International Double-Blind Actovegin): A Randomized Controlled Trial to Assess the Efficacy of Actovegin in Poststroke Cognitive Impairment. Stroke. 2017 May;48(5):1262-1270. doi: 10.1161/STROKEAHA.116.014321. PMID 28432265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 33 investigative sites in Belarus, Kazakhstan and Russia from 28 June 2012 to 26 November 2014.
Pre-assignment Details: Participants who had suffered ischaemic stroke were enrolled equally in 1 of 2 treatment groups, actovegin 2000 mg solution (up to 20 infusions) followed by 200 mg tablets 3 times a day or placebo.
Period: Overall Study
Arm/Group | Actovegin | Placebo
Started | 248 | 255
Completed | 212 | 221
Not Completed | 36 | 34
Not completed — Death | 8 | 5
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Participant | 8 | 11
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Recurrent Stroke | 13 | 8
Not completed — Disallowed Concomitant Medication | 3 | 2
Not completed — Carotid or Neurosurgery | 0 | 1
Not completed — General Anaesthesia | 0 | 1
Not completed — Other Miscellaneous Reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Actovegin | Placebo | Total
Number analyzed (Participants) | 248 | 255 | 503
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (6.65) | 69.6 (7.18) | 69.9 (6.92)
Age, Customized [Number; unit: participants]
  ≤ 65 years | 78 | 97 | 175
  > 65 years | 170 | 158 | 328
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 142 | 262
  Male | 128 | 113 | 241
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 3 | 6
  Black or African American | 1 | 1 | 2
  White | 240 | 248 | 488
  Other | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Russia | 190 | 195 | 385
  Kazakhstan | 2 | 2 | 4
  Belarus | 56 | 58 | 114
Height [Mean (Standard Deviation); unit: cm] | 167.6 (7.47) | 167.2 (7.89) | 167.4 (7.68)
Weight [Mean (Standard Deviation); unit: kg] | 78.3 (13.76) | 78.0 (13.73) | 78.1 (13.73)
Number of Years of Education [Mean (Standard Deviation); unit: years] | 12.2 (3.41) | 12.3 (3.40) | 12.3 (3.40)
Diabetes [Number; unit: participants]
  Yes | 40 | 57 | 97
  No | 208 | 198 | 406
Ischaemic Heart Disease or Peripheral Artery Disease [Number; unit: participants]
  Yes | 245 | 253 | 498
  No | 3 | 2 | 5
Previous Ischaemic Stroke [Number; unit: participants]
  Yes | 40 | 38 | 78
  No | 208 | 217 | 425
Smoking Status [Number; unit: participants]
  Never smoked | 172 | 195 | 367
  Current smoker | 53 | 37 | 90
  Ex-smoker | 23 | 23 | 46
Alcohol Consumption [Number; unit: participants]
  Never drank | 117 | 126 | 243
  Occasional drinker | 131 | 128 | 259
  Daily drinker | 0 | 1 | 1
Fertility Status of Female Participants [Number; unit: participants] — Female participants with available fertility status data only: 120 and 142 participants in each treatment arm, respectively.
  participants
    Surgically Sterile/Hysterectomized | 3 | 5 | 8
    Post-menopausal | 117 | 137 | 254

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale + Cognitive Subscale Extended Version (ADAS-cog+) at Month 6
Description: The ADAS-cog measures cognitive performance by combining the ratings of 11 items. The cognitive domains mainly addressed by ADAS-cog are: memory (short term), language, ability to orientate (reflects memory), construction/planning of simple designs and performance. The extended version of the ADAS-cog (ADAS-cog+) includes 3 additional items: a 2-number cancellation task to test for attention, a delayed recall task to test for memory consolidation and a maze test for executive performance. Each item is scored and then the item scores are totaled. Total scores range from 0 (best) to 90 (worst). Higher scores indicate greater cognitive impairment. A negative change from Baseline indicates improvement.
  Analysis of Covariance (ANCOVA) model was used for analyses that included treatment, pooled centre, and their interaction as factors and Baseline ADAS-cog+ score as a covariate.
Time Frame: Baseline and Month 6
Population: Intent-to-treat population, all enrolled participants who received at least one dose of study drug, with data available for analysis. Missing individual item scores (where only some item scores missing) imputed with worst possible score and missing total scores (where all item scores missing) imputed by last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 224 | 234
score on a scale | -6.8 (0.58) | -4.6 (0.58)
Statistical Analysis 1: Comparison: Actovegin vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -2.3, 95% CI 2-sided [-3.9 to -0.7], Standard Error of Mean 0.82

2. Secondary Outcome: Change From Baseline in ADAS-cog+ at Month 3 and Month 12
Description: The ADAS-cog measures cognitive performance by combining the ratings of 11 items. The cognitive domains mainly addressed by ADAS-cog are: memory (short term), language, ability to orientate (reflects memory), construction/planning of simple designs and performance. The extended version of the ADAS-cog (ADAS-cog+) includes 3 additional items: a 2-number cancellation task to test for attention, a delayed recall task to test for memory consolidation and a maze test for executive performance. Each item is scored and then the item scores are totaled. Total scores range from 0 (best) to 90 (worst). Higher scores indicate greater cognitive impairment. A negative change from Baseline indicates improvement.
  ANCOVA model was used for analyses that included treatment, pooled centre, and their interaction as factors and Baseline ADAS-cog+ score as a covariate.
Time Frame: Baseline and Months 3 and 12
Population: Intent-to-treat population, all enrolled participants who received at least one dose of study drug, with data available for analysis. Missing individual item scores (where only some item scores missing) imputed with worst possible score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
score on a scale
  Change from Baseline at Month 3 (n=224, 234) | -5.4 (0.53) | -4.3 (0.52)
  Change from Baseline at Month 12 (n=211, 219) | -8.2 (0.66) | -4.5 (0.66)
Statistical Analysis 1: Comparison: Actovegin vs Placebo; Month 3; Test type: Superiority or Other; p = 0.122, ANCOVA; LS Mean Difference = -1.1, 95% CI 2-sided [-2.6 to 0.3], Standard Error of Mean 0.74
Statistical Analysis 2: Comparison: Actovegin vs Placebo; Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -3.7, 95% CI 2-sided [-5.5 to -1.9], Standard Error of Mean 0.93

3. Secondary Outcome: Change From Baseline in Montreal Cognitive Assessment Scale (MoCA) at End of Infusion Period, Months 3, 6 and 12
Description: The MoCA is a rapid screening test to assess mild cognitive impairment. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 0 to 30 points; a score of 26 or above is considered normal. A positive change from Baseline (BL) indicates improvement.
  ANCOVA model was used for analyses that included treatment and pooled centres as factors, plus years of education and baseline MoCA score as covariates.
Time Frame: Baseline, End of Infusion and Months 3, 6 and 12
Population: Participants from the Intent-to-treat population, all enrolled participants who received at least one dose of study drug, with data available for analyses at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
score on a scale
  Change from BL at End of Infusion (n=242, 247) | 2.1 (0.15) | 1.8 (0.15)
  Change from Baseline at Month 3 (n=224, 234) | 3.4 (0.20) | 2.7 (0.20)
  Change from Baseline at Month 6 (n=217, 228) | 3.8 (0.21) | 3.1 (0.21)
  Change from Baseline at Month 12 (n=211, 220) | 3.9 (0.25) | 2.9 (0.24)
Statistical Analysis 1: Comparison: Actovegin vs Placebo; End of Infusion Period; Test type: Superiority or Other; p = 0.111, ANCOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Actovegin vs Placebo; Month 3; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = 0.7, 95% CI 2-sided [0.1 to 1.2], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Actovegin vs Placebo; Month 6; Test type: Superiority or Other; p = 0.013, ANCOVA; LS Mean Difference = 0.7, 95% CI 2-sided [0.2 to 1.3], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Actovegin vs Placebo; Month 12; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = 1.0, 95% CI 2-sided [0.3 to 1.7], Standard Error of Mean 0.34

4. Secondary Outcome: Percentage of ADAS-cog+ Responders at Time Points 3, 6 and 12 Months
Description: Responder was defined as an improvement of 4 or more from baseline on the ADAS-cog+ scale using observed data. The proportion of responders was compared between treatments using a chi-square test.
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 3
Measure: Number; unit: percentage of responders
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
percentage of responders
  Month 3 (n=215, 223) | 59.1 | 48.9
  Month 6 (n=208, 216) | 62.5 | 52.3
  Month 12 (n=200, 207) | 69.0 | 58.9
Statistical Analysis 1: Comparison: Actovegin vs Placebo; Month 3; Test type: Superiority or Other; p = 0.032, Chi-squared; Percent Difference = 10.2, 95% CI 2-sided [0.9 to 19.5]
Statistical Analysis 2: Comparison: Actovegin vs Placebo; Month 6; Test type: Superiority or Other; p = 0.034, Chi-squared; Percent Difference = 10.2, 95% CI 2-sided [0.8 to 19.5]
Statistical Analysis 3: Comparison: Actovegin vs Placebo; Month 12; Test type: Superiority or Other; p = 0.035, Chi-squared; Percent Difference = 10.1, 95% CI 2-sided [0.8 to 19.3]

5. Secondary Outcome: Percentage of Participants With a Diagnosis of Dementia
Description: Diagnosis of dementia will be evaluated after 6 and 12 months classified according to International Statistical Classification of Diseases and related Health Problems 10th Revision (ICD-10) [Classification of Mental and Behavioural Disorders, Diagnostic Criteria for Research]. The proportion of participants with dementia was compared between treatments using a Fisher's exact test.
Time Frame: Month 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 218 | 228
percentage of participants
  Month 6 | 7.3 | 10.5
  Month 12 | 8.7 | 12.7
Statistical Analysis 1: Comparison: Actovegin vs Placebo; Month 6; Test type: Superiority or Other; p = 0.251, Fisher Exact; Percent Difference = -3.2, 95% CI 2-sided [-8.5 to 2.1]
Statistical Analysis 2: Comparison: Actovegin vs Placebo; Month 12; Test type: Superiority or Other; p = 0.221, Fisher Exact; Percent Difference = -4.0, 95% CI 2-sided [-9.7 to 1.7]

6. Secondary Outcome: Change From Baseline in National Institutes of Health Stroke Scale (NIHSS) at End of Infusion Period, Months 3, 6 and 12
Description: The NIHSS is a tool to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 (normal) to 4 (some level of impairment). The individual scores from each item are summed in order to calculate total possible NIHSS score from 0 (best) to 42 (worst). A negative change from Baseline indicates improvement. ANCOVA model was used for analyses that included treatment and pooled centre as factors and Baseline NIHSS score as a covariate.
Time Frame: Baseline and End of Infusion and Months 3, 6 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
score on a scale
  Change from BL at End of Infusion (n=243, 248) | -1.8 (0.10) | -1.7 (0.10)
  Change from Baseline at Month 3 (n=224, 235) | -2.9 (0.10) | -2.7 (0.10)
  Change from Baseline at Month 6 (n=219, 228) | -3.2 (0.10) | -3.2 (0.10)
  Change from Baseline at Month 12 (n=211, 220) | -3.5 (0.10) | -3.4 (0.10)
Statistical Analysis 1: Comparison: Actovegin vs Placebo; End of Infusion Period; Test type: Superiority or Other; p = 0.239, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Actovegin vs Placebo; Month 3; Test type: Superiority or Other; p = 0.136, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Actovegin vs Placebo; Month 6; Test type: Superiority or Other; p = 0.890, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Actovegin vs Placebo; Month 12; Test type: Superiority or Other; p = 0.455, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14

7. Secondary Outcome: Barthel Index at Months 3 and 6
Description: The Barthel Index consists of 10 items that measure a person's daily functioning, specifically the activities of daily living and mobility. The items include: feeding, transfers (bed to chair and back), grooming, toilet use, bathing, mobility (walking on level surface), going up and down stairs, dressing, continence of bowels and bladder. Each performance item is rated, with a given number of points assigned to each level or ranking. Individual scores are summed for a total possible scores ranging from 0 (worst) to 100 (best) with higher scores indicating more independent daily living.
Time Frame: Months 3 and 6
Population: as for outcome 3
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
score on a scale
  Month 3 (n=224,235) | 100.0 [55.0 to 100.0] | 100.0 [9.0 to 100.0]
  Month 6 (n=219,228) | 100.0 [55.0 to 100.0] | 100.0 [50.0 to 100.0]

8. Secondary Outcome: EuroQol EQ-5D (EQ-5D) at Month 6
Description: EQ-5D is a standardized measure of health status consisting of 5 dimensions: mobility, self -care, usual activities, pain/discomfort and anxiety/depression. The participant rates their level of function in each area using a 5 point scale where 1=no problems (best) to 5=extreme problems (worst). The percentage of participants in each category is reported.
Time Frame: Month 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 219 | 224
percentage of participants
  Mobility_No problem | 41.5 | 32.2
  Mobility_Slight problem | 29.8 | 31.8
  Mobility_Moderate problem | 12.5 | 16.5
  Mobility_Severe problem | 4.0 | 7.1
  Mobility_Unable | 0.4 | 0.4
  Self-care_No problem | 58.5 | 48.6
  Self-care_Slight problem | 19.8 | 25.5
  Self-care_Moderate problem | 7.7 | 9.8
  Self-care_Severe problem | 2.0 | 3.5
  Self-care_Unable | 0.4 | 0.4
  Usual activities_No problem | 32.7 | 32.9
  Usual activities_Slight problem | 40.7 | 34.5
  Usual activities_Moderate problem | 8.9 | 17.3
  Usual activities_Severe problem | 4.0 | 2.5
  Usual activities_Unable | 2.0 | 0.8
  Pain or discomfort_No pain | 50.0 | 46.3
  Pain or discomfort_Slight pain | 30.6 | 25.5
  Pain or discomfort_Moderate pain | 6.0 | 15.3
  Pain or discomfort_Severe pain | 0.8 | 0.8
  Pain or discomfort_Extreme pain | 0.4 | 0
  Anxiety or depression_Not anxious | 50.0 | 48.2
  Anxiety or depression_Slightly anxious | 31.0 | 29.4
  Anxiety or depression_Moderately anxious | 6.0 | 9.4
  Anxiety or depression_Severely anxious | 0.8 | 0.8
  Anxiety or depression_Extremely anxious | 0.4 | 0

9. Secondary Outcome: EuroQol EQ-5D (EQ-5D) at Month 12
Description: as for outcome 8
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 212 | 220
percentage of participants
  Mobility_No problem | 37.9 | 36.5
  Mobility_Slight problem | 31.0 | 29.4
  Mobility_Moderate problem | 12.5 | 11.8
  Mobility_Severe problem | 3.2 | 7.5
  Mobility_Unable | 0.8 | 0.8
  Self-care_No problem | 55.2 | 48.2
  Self-care_Slight problem | 22.2 | 23.5
  Self-care_Moderate problem | 6.0 | 9.4
  Self-care_Severe problem | 1.6 | 3.9
  Self-care_Unable | 0.4 | 0.8
  Usual activities_No problem | 32.7 | 31.0
  Usual activities_Slight problem | 39.1 | 33.7
  Usual activities_Moderate problem | 9.7 | 15.7
  Usual activities_Severe problem | 2.8 | 4.3
  Usual activities_Unable | 1.2 | 1.2
  Pain or discomfort_No pain | 46.8 | 46.7
  Pain or discomfort_Slight pain | 28.6 | 26.3
  Pain or discomfort_Moderate pain | 8.5 | 11.4
  Pain or discomfort_Severe pain | 1.6 | 1.2
  Pain or discomfort_Extreme pain | 0 | 0.4
  Anxiety or depression_Not anxious | 48.4 | 47.1
  Anxiety or depression_Slightly anxious | 31.5 | 27.1
  Anxiety or depression_Moderately anxious | 4.8 | 10.6
  Anxiety or depression_Severely anxious | 0.8 | 0.8
  Anxiety or depression_Extremely anxious | 0 | 0.4

10. Secondary Outcome: EuroQol EQ-5D (EQ-5D) General Health at Months 6 and 12
Description: The EuroQoL included a visual analogue scale where the subject marks how they feel at that moment on a scale from 0 (the worst health that can be imagined) to 100 (the best health that can be imagined).
Time Frame: Months 6 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
score on a scale
  Month 6 (n=219, 224) | 67.3 (16.04) | 65.0 (16.82)
  Month 12 (n=212, 220) | 67.8 (15.87) | 65.6 (17.51)

11. Secondary Outcome: Beck Depression Inventory, Version II (BDI-II) at Months 3, 6 and 12
Description: The BDI-II is a 21-question multiple-choice self-report inventory for measuring the severity of depression. is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex. Each answer is scored on a scale 0 (best) to 3 (worst). Total scores range from 0 to 63 with higher scores indicating more severe depression.
  BDI II scale:
  * 0-13 minimal depression
  * 14-19 mild depression
  * 20-28 moderate depression
  * 29-63 severe depression
Time Frame: Months 3, 6 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
score on a scale
  Month 3 (n=224, 234) | 12.5 (11.02) | 11.6 (8.08)
  Month 6 (n=219, 227) | 11.3 (8.88) | 11.5 (10.58)
  Month 12 (n=212, 220) | 10.7 (7.10) | 11.5 (8.24)

12. Secondary Outcome: Percentage of Participants With a Diagnosis of Dementia
Description: Diagnosis of dementia will be evaluated after 6 and 12 months classified according to International Statistical Classification of Diseases and related Health Problems 10th Revision (ICD-10) [Classification of Mental and Behavioural Disorders, Diagnostic Criteria for Research].
Time Frame: Month 6 and 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Actovegin | Placebo
Number analyzed (Participants) | 248 | 255
percentage of participants
  Month 6 | 7.3 | 10.5
  Month 12 | 8.7 | 12.7

ADVERSE EVENTS:
Time Frame: First dose of study drug to 10 days after last dose of study drug (up to approximately 6.5 months).
Description: Any adverse events and abnormal laboratory findings irrespective of the relation to study treatment were documented. Safety population included all participants who received at least 1 dose of study drug based on treatment received. 2 participants in the placebo arm received actovegin and are included in the actovegin arm for safety analyses.
Arm/Group | Actovegin | Placebo
Serious Adverse Events (participants affected / at risk) | 22/250 | 17/253
Other Adverse Events (participants affected / at risk) | 31/250 | 31/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Actovegin (N=250) | Placebo (N=253)
Ischaemic stroke (Nervous system disorders) | 13 | 5 — One treatment-emergent death occurred during treatment with actovegin and is not related and two treatment-emergent deaths occurred during treatment with placebo (1 of which also had Brain oedema and Hypostatic pneumonia) and are not related.
Brain oedema (Nervous system disorders) | 1 | 2 — One treatment-emergent death occurred during treatment with actovegin and is not related and two treatment-emergent deaths occurred during treatment with placebo (1 participant also had Ischaemic stroke and Hypostatic pneumonia) and are not related.
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with actovegin and is not related.
Cerebrovascular accident (Nervous system disorders) | 0 | 1
VIIth Nerve Paralysis (Nervous system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 — One treatment-emergent death occurred during treatment with actovegin and is not related.
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with actovegin and is not related.
Coronary artery disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1 — One treatment-emergent death occurred during treatment with placebo and is not related.
Pneumonia (Infections and infestations) | 1 | 0 — One treatment-emergent death occurred during treatment with actovegin and is not related.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Two treatment-emergent deaths occurred during treatment with actovegin and are not related.
Arteriosclerosis (Vascular disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with placebo and is not related.
Hypertensive crisis (Vascular disorders) | 1 | 0
Death (General disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with placebo and is not related. No specific cause of death was identified or reported by the investigator.
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Actovegin (N=250) | Placebo (N=253)
Atrial fibrillation (Cardiac disorders) | 5 | 3
Respiratory tract infection viral (Infections and infestations) | 5 | 8
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 2
Amnesia (Nervous system disorders) | 0 | 7
Dementia (Nervous system disorders) | 5 | 9
Headache (Nervous system disorders) | 7 | 7
Hypertension (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.